CLINICAL TRIAL: NCT00565422
Title: Efficacy of Escitalopram in the Treatment of Internet Addiction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Dr. Eric Hollander, Mount Sinai School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXP-MD-09; 01-1174
Record Dates: First submitted 2007-11-28; First posted 2007-11-30 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Internet Addiction
Keywords: Internet addiction; Problematic internet use; Escitalopram; Lexapro
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Escitalopram
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — 10 mg/day
  Other Names: Lexapro

SUMMARY:
The purpose of this study was to determine whether Lexapro (Escitalopram) is safe and effective in treating problematic internet use.

DETAILED DESCRIPTION:
Many individuals experience marked distress and functional impairments as a result of their perceived inability to control their 'non-essential' (non-job/school related) use of the Internet. Frequently these people develop a preoccupation with the Internet, a need for escape to the Internet, and increasing irritability when trying to cut back use of the Internet. There have been no studies to date looking at the effectiveness of medications in the treatment of this disorder. In our clinical experience, we find these patients with Internet addiction usually respond to serotonin reuptake inhibitors within 12 weeks. This study will examine the efficacy of escitalopram in Internet addiction among adults.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed an informed consent form
2. Current diagnosis of Internet addiction
3. Age ³ 18
4. Subject must be able to take oral medication
5. Subject may be in psychotherapy initiated at least three months prior to Screening. Subject must not discontinue or otherwise alter this therapy during the study.
6. In the opinion of the investigator, the subject is capable of complying with all study procedures.

Exclusion Criteria:

1. Current suicidal or homicidal ideation
2. Subject has a primary diagnosis of schizophrenia or other psychotic disorders
3. Subject has a primary diagnosis of Bipolar I disorder
4. Current pedophilia
5. Current DSM-IV diagnosis of substance dependence or abuse, excluding nicotine
6. Women of child-bearing potential who are pregnant, nursing, or not using contraception
7. Use of antidepressants at a therapeutic level for the treatment of problematic internet use within 2 weeks prior to study entry (or 4 weeks for use of MAOIs, or 6 weeks for use of fluoxetine)
8. Current use of antidepressants at a therapeutic level for the treatment of a disorder other than problematic internet use
9. Subject has any organic mental disorder
10. Clinically significant unstable medical disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2002-12; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
length of non-essential Internet use in hours/week as well as CGI-Improvement | baseline and biweekly for 10 weeks

SECONDARY OUTCOMES:
ratings on depression, anxiety, impulsivity, self-esteem, obsessive-compulsive symptoms | baseline and biweekly for 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai

REFERENCES:
- [Derived] Dell'Osso B, Hadley S, Allen A, Baker B, Chaplin WF, Hollander E. Escitalopram in the treatment of impulsive-compulsive internet usage disorder: an open-label trial followed by a double-blind discontinuation phase. J Clin Psychiatry. 2008 Mar;69(3):452-6. doi: 10.4088/jcp.v69n0316. PMID 18312057